CLINICAL TRIAL: NCT00209014
Title: Phase II Trial of Thalidomide in Refractory/Relapsed Diffuse Large B-Cell Lymphoma and Hodgkin's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Celgene unable to continue funds.
Sponsor: Emory University (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Leonard Heffner, MD, Emory University Winship Cancer Institute
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0544-2003
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2009-05-07 (Estimated); Status verified 2009-05

CONDITIONS: B-Cell Lymphoma; Hodgkin's Disease
Keywords: B-Cell Lymphoma; Hodgkin's Disease
MeSH Terms: conditions — Lymphoma, B-Cell; Hodgkin Disease | interventions — Thalidomide

INTERVENTIONS:
Drug: Thalidomide

SUMMARY:
Patients who have relapsed or refractory large B-cell lymphoma are being asked to take part in this study. The purpose of this study is to find out what effects (good and bad) the drug thalidomide has on patients and the lymphoma.

DETAILED DESCRIPTION:
Patients who have relapsed or refractory large B-cell lymphoma are being asked to take part in this study. This research is being done because current treatment does not help everyone with this disease. The purpose of this study is to find out what effects (good and bad) the drug thalidomide has on patients and the lymphoma. Thalidomide has been shown to have activity against other cancers but is not approved by the FDA for treatment of lymphoma. Thalidomide prevents growth of new blood vessels that allow cancer cells to receive nourishment and spread. Another reason for doing the study is that researchers want to learn more about how the drug works and whether some patients respond better than others.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an expected survival period of 6 months or greater and who have been diagnosed with any stage of diffuse large B-cell lymphoma or Hodgkin's disease will be eligible to participate in this study. Final eligibility will be determined by the health professionals conducting this trial.

Exclusion Criteria:

* Women who are pregnant, lactating or who refuse to have a pregnancy test will not be eligible for this study. Also, patients with an active infection, or a history of current or previous deep vein thrombosis and/or currently receiving anticoagulant therapy for deep vein thrombosis will be excluded from participation in this study. Final eligibility will be determined by the health professionals conducting this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2003-07; Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: L. Thompson Heffner, MD, Principal Investigator — Emory University Winship Cancer Institute
Locations (1):
- Emory University Winship Cancer Institute, Atlanta, Georgia, United States